CLINICAL TRIAL: NCT05974176
Title: Evaluating the Effectiveness of Evidence-based Trauma Interventions (Trauma Focused CBT - TF-CBT; and Trauma Systems Therapy - TST), Baseline Index Trauma, and PTSD Symptoms in the Context of Contributing Stress From Racialized Trauma and Acculturation Stress
Brief Title: Considering Racial and Acculturation Stress in Addressing Trauma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-00094
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Trauma-related PTSD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trauma Focused CBT (TF-CBT) (Experimental): Patients and families randomized to engage in TF-CBT.
  Interventions: Behavioral: Trauma Focused CBT (TF-CBT)
- Trauma Systems therapy (TST) (Experimental): Patients and families randomized to engage in TST.
  Interventions: Behavioral: Trauma Systems therapy (TST)

INTERVENTIONS:
Behavioral: Trauma Focused CBT (TF-CBT) — TF-CBT is an evidence-based treatment for children and adolescents impacted by trauma and their parents or caregivers. It is a components-based treatment model that incorporates trauma-sensitive interventions with cognitive behavioral, family, and humanistic principles and techniques.
  Arms: Trauma Focused CBT (TF-CBT)
Behavioral: Trauma Systems therapy (TST) — Trauma Systems Therapy (TST) is focused on the factors that contribute to children and adolescents who experience traumatic stress through the lens of the social context, vulnerabilities, and strengths of the person undergoing treatment.
  Arms: Trauma Systems therapy (TST)

SUMMARY:
Investigators plan to offer two evidence based interventions - Trauma Focused Cognitive Behavioral Therapy (CBT) (TF-CBT) and Trauma Systems therapy (TST) to traumatized children and their families. The investigators are looking to evaluate the effectiveness of these interventions in the context of additional stress related to racialized trauma and acculturation stress

ELIGIBILITY:
Inclusion Criteria:

* Child/adolescent aged 5-17 years of age who has experienced trauma with associated and related emotional dysregulation (i.e PTSD) and one of their parent/guardian
* Have capacity and willingness to provide consent or age-appropriate assent

Exclusion Criteria:

* Individual with intellectual disability with an IQ<70
* Individual with active suicidality, homicidality, or other symptoms at the time of enrollment that warrants hospitalization

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 237 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Child and Adolescent Trauma Screen (CATS) Score at Baseline | Baseline (Day 1)
  CATS is a 15-item assessment of potentially traumatic events and of posttraumatic stress symptoms. The total score is the sum of responses and ranges from 0-60; higher scores indicates more symptoms.
CATS Score at Completion of Intervention | Completion of Intervention (Typically Month 3-4)
  CATS is a 15-item assessment of potentially traumatic events and of posttraumatic stress symptoms. The total score is the sum of responses and ranges from 0-60; higher scores indicates more symptoms.

SECONDARY OUTCOMES:
Acculturative Stress Scale (SAFE) Score at Baseline | Baseline (Day 1)
  SAFE is a 24-item assessment of acculturative stress. Items are rated on a scale from 1 (not at all true) to 4 (very true). The total score is the sum of responses and ranges from 24 to 96; higher scores indicate greater levels of acculturative stress.
SAFE Score at Completion of Intervention | Completion of Intervention (Typically Month 3-4)
  SAFE is a 24-item assessment of acculturative stress. Items are rated on a scale from 1 (not at all true) to 4 (very true). The total score is the sum of responses and ranges from 24 to 96; higher scores indicate greater levels of acculturative stress.
Bidimensional Acculturation Scale (BAS) Score at Baseline | Baseline (Day 1)
  BAS is a 24-item assessment of bidimensional acculturation. Items are rated on a 4-point scale. The total score is the sum of responses and ranges from 24 to 96; higher scores indicate higher levels of bidimensional acculturation.
BAS Score at Completion of Intervention | Completion of Intervention (Typically Month 3-4)
  BAS is a 24-item assessment of bidimensional acculturation. Items are rated on a 4-point scale. The total score is the sum of responses and ranges from 24 to 96; higher scores indicate higher levels of bidimensional acculturation.
Multi-Group Ethnic Identity Measure (MEIM-6) Score at Baseline | Baseline (Day 1)
  6-item questionnaire to assess the degree of ethnic identity among adolescents. Each item is rated on a scale from 1 (strongly disagree) to 5 (strongly agree). The total score is the sum of responses and ranges from 6 to 30; higher scores indicate greater ethnic identify.
Multi-Group Ethnic Identity Measure (MEIM-6) Score at Completion of Intervention | Completion of Intervention (Typically Month 3-4)
  6-item questionnaire to assess the degree of ethnic identity among adolescents. Each item is rated on a scale from 1 (strongly disagree) to 5 (strongly agree). The total score is the sum of responses and ranges from 6 to 30; higher scores indicate greater ethnic identify.
Trauma Symptoms of Discrimination Scale (TSDS) at Baseline | Baseline (Day 1)
  21-item questionnaire assessing trauma symptoms of discrimination. Each item is rated on a scale from 1 (never) to 4 (often). The total score is the sum of responses and ranges from 21 to 84; higher scores indicate greater symptoms.
Trauma Symptoms of Discrimination Scale (TSDS) at Completion of Intervention | Completion of Intervention (Typically Month 3-4)
  21-item questionnaire assessing trauma symptoms of discrimination. Each item is rated on a scale from 1 (never) to 4 (often). The total score is the sum of responses and ranges from 21 to 84; higher scores indicate greater symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Reliford, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Shared only with study team.